CLINICAL TRIAL: NCT04838158
Title: Assessment of Knee Flexor Muscles Strength in Patients With Patellar Instability and Its Clinical Implication in Non-surgical Treatment of Patients After First Patella Dislocation.
Brief Title: Assessment of Knee Flexor Muscles Strength in Patients With Patellar Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PolishMMHRI 23/06/2010
Record Dates: First submitted 2021-03-22; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-01

CONDITIONS: Patella Dislocation Recurrent; Children, Only

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Those cases who underwent operative treatment and isokinetics evaluation.
  Interventions: Diagnostic Test: Isokinetic measurements
- Control group (Other): Those who were control group of healthy subjects to compare to normative data
  Interventions: Diagnostic Test: Isokinetic measurements

INTERVENTIONS:
Diagnostic Test: Isokinetic measurements — Each patient underwent an isokinetic examination on Biodex System 3 (Biodex Multi-Joint System - Pro, Biodex Medical Systems, Inc. New York, USA). In the study group, both side hamstring muscle were evaluated at the velocities of 60 and180 deg/s for the following parameters: peak torque (PT), torque in 30 degree of the knee flexion (T 30 deg.), angle of peak torque (APT) and peak torque hamstring to quadriceps ratio (H/Q ratio).

SUMMARY:
The study enrolled 33 patients with confirmed recurrent patellar dislocation, including 6 patients with bilateral involvement. In the study group, both side hamstring muscle were evaluated at the velocities of 60 and 180 deg/s for the following parameters: peak torque, torque in 30 degree of the knee flexion, angle of peak torque and peak torque hamstring to quadriceps ratio (H/Q ratio).

DETAILED DESCRIPTION:
The study enrolled 33 patients with confirmed recurrent patellar dislocation, including 6 patients with bilateral involvement. The study group consisted of 20 girls and 13 boys with average age at the time of the study 16.2 years (range: 8 to 17 years, SD 2.7). For the purpose of the study, a control group of 18 healthy subjects (12 girls and 6 boys) aged on the average 15.7 years (range:13 to 17 years, SD 1.5), was recruited.

The following study inclusion criteria were applied: recurrent patellar dislocation, correctly completed testing protocol, age under 18 years at the time of testing. Subjects with osteochondral fracture and those with a history of the knee surgery were excluded.

Each patient underwent an isokinetic examination on Biodex System 3 (Biodex Multi-Joint System - Pro, Biodex Medical Systems, Inc. New York, USA). In the study group, both side hamstring muscle were evaluated at the velocities of 60 and180 deg/s for the following parameters: peak torque (PT), torque in 30 degree of the knee flexion (T 30 deg.), angle of peak torque (APT) and peak torque hamstring to quadriceps ratio (H/Q ratio).

Isokinetic measurements were made by a trained, experienced physiotherapist. After a proper warm-up and instruction, the test performed 10 full repetitions, the best result was recorded. The results of the peak torque (PT) of both test and control limbs were then compared with the normative data for age and gender available in the literature. In addition, we compared the peak torque (PT), torque in 30 degrees of the knee flexion (T 30 deg.), angle of peak torque (APT) and peak torque hamstring to quadriceps ratio (H/Q ratio) of involved and uninvolved knee flexor strength in the study group. Depending on the data distribution, the nonparametric Wilcoxon's test or the parametric t-test for the related data was applied. Statistical significance was assumed for p<0.05. The study was approved by our Institutional Review Board. Informed consent was obtained and the rights of subjects were protected.

ELIGIBILITY:
Inclusion Criteria:

* recurrent patellar dislocation,
* correctly completed testing protocol,
* age under 18 years at the time of testing

Exclusion Criteria:

* osteochondral fracture
* those with a history of the knee surgery

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2016-01-30 (Actual)

PRIMARY OUTCOMES:
hamstrings peak torque | up to 18 months
  measured on Biodex System
torque in 30 degrees of the knee flexion | up to 18 months
  measured on Biodex System
angle of peak torque | up to 18 months
  measured on Biodex System
peak torque hamstring to quadriceps ratio (H/Q ratio) | up to 18 months
  measured on Biodex System

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Małecki, Ph.D., Study Director — Polish Mother's Memorial Hospital Research Institute; Jarosław Fabiś, prof., Study Chair — Medical University of Lodz; Paweł Flont, Ph.D., Principal Investigator — Polish Mother's Memorial Hospital Research Institute; Anna Fabiś-Strobin, Ph.D., Principal Investigator — Polish Mother's Memorial Hospital Research Institute; Kryspin Niedzielski, prof., Study Chair — Polish Mother's Memorial Hospital Research Institute

IPD SHARING:
Plan to Share IPD: Yes
Research protocol, personal results, informed consent
Supporting Information: Study Protocol, ICF
Time Frame: April 2021 - December 2023
Access Criteria: Upon reasonable request on e-mail krzynormal@wp.pl

REFERENCES:
- [Derived] Malecki K, Fabis J, Flont P, Fabis-Strobin A, Niedzielski K. Assessment of knee flexor muscles strength in patients with patellar instability and its clinical implications for the non-surgical treatment of patients after first patellar dislocation - pilot study. BMC Musculoskelet Disord. 2021 Aug 28;22(1):740. doi: 10.1186/s12891-021-04636-4. PMID 34454460